CLINICAL TRIAL: NCT03288519
Title: The Use of the Classic Laryngeal Mask Airway in Patients With Cerebral Aneurysm Undergoing Endovascular Therapy
Brief Title: Use of Classic LMA During Endovascular Therapy
Status: Completed | Type: Observational
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2017-08-31; First posted 2017-09-20 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2017-09

CONDITIONS: Cerebral Aneurysm Unruptured; Cerebral Aneurysm; Hemodynamic Instability; Airway Morbidity
Keywords: Cerebral aneurysm; Endovascular therapy; Classic laryngeal mask airway; Hemodynamic changes
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Earlier treatment and resolution for patients with cerebral aneurysms is now possible due to earlier diagnosis. This observational study aims to evaluate the intraoperative cardiovascular parameters in patients with cerebral aneurysms undergoing endovascular therapy.

Method: This is an observational prospective study. Patients ≥ 18 years old diagnosed with an unruptured cerebral aneurysm or subarachnoid hemorrhage (SAH) (Hunt & Hess grade I or II) undergoing endovascular treatment under general anesthesia between April 2015 and February 2017 were included. Non-invasive measurements of hemodynamic variables were collected at six time points during the procedure (T1 to T6). Statistical analysis was performed by using central tendency measures for quantitative variables and absolute / relative frequency measurements for qualitative variables.

DETAILED DESCRIPTION:
Objective

• To assess the usefulness of general anesthesia with Laryngeal Mask Airway (LMA)-Classic for the endovascular treatment of cerebral aneurysms based on cardiovascular stability analysis Data collection Anesthetic protocol was standardized for all patients consisting of an intravenous induction with fentanyl (1-2 μg/kg), lidocaine (1.5 mg/kg), propofol (2 mg/kg), and dexamethasone (8 mg) followed by the insertion of the LMA-Classic. Sevoflurane with a minimal alveolar concentration (MAC) between 0.9 and 1.1%, dipyrone (2 gr IV), and morphine (0.05 mg/kg IV) were used during maintenance. Tidal volume (VT) and respiratory rate (RR) were adjusted to 7 ml/Kg and 12-14 per minute respectively. Non-invasive hemodynamic monitoring included mean arterial pressure (MAP), heart rate (HR), oxygen saturation, and end-tidal carbon dioxide (ETCO2).

Data was collected within six time points: Time point 1: before induction, Time point 2: after induction, Time point 3: after LMA-Classic insertion, Time point 4: during the endovascular procedure, Time point 5: during coiling, and Time point 6: at the end of the procedure and LMA-Classic removal.

The following demographic and clinical data were collected: age, gender, American Society of Anesthesiologists Physical Status (ASA-PS), total procedure time, comorbidities, aneurysm location, and associated clinical manifestations. Adverse events, such as intraoperative aneurysm rupture or need for endotracheal intubation, will be recorded.

Ethical considerations Approvals were obtained from the ethics committees at Antioquia University and Especialidades Médicas Metropolitanas Sociedad Anónima (EMMSA) Clinic. Patients signed an informed consent and confidentiality agreement before participating.

Statistical analysis Data was collected in an excel spreadsheet (Microsoft Excel 2010®), SAS 9.4 (SAS Institute, Cary, N.C.) was used for subsequent analysis. Continuous variables were summarized as means and standard deviations (SD). Categorical variables were summarized as frequencies and percentages. Linear mixed models were fit to model continuous clinical variables over time using contrasts to test differences between time points. P-values less than 0.05 were considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Diagnosed with an unruptured cerebral aneurysm or SAH (Hunt & Hess grade I or II)
* Planned to undergo endovascular therapy under general anesthesia between April 2015 and February 2017 in the Especialidades Médicas Metropolitanas Sociedad Anónima (EMMSA) Clinic in Bello, Antioquia, Colombia

Exclusion Criteria:

* Patients diagnosed with a cerebral aneurysm undergoing craniotomy and clipping and patients with SAH (Hunt & Hess grade > II).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An observational prospective study was undertaken in the Especialidades Médicas Metropolitanas Sociedad Anónima (EMMSA) Clinic in Bello, Antioquia, Colombia. The investigators included patients ≥ 18 years old diagnosed with an unruptured cerebral aneurysm or SAH (Hunt & Hess grade I or II) undergoing endovascular treatment under general anesthesia between April 2015 and February 2017. The investigators excluded patients diagnosed with a cerebral aneurysm undergoing craniotomy and clipping and patients with SAH (Hunt & Hess grade > II).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Hemodynamic changes (changes from baseline in Heart Rate and Mean Arterial Pressure) | Outcome measure will be assessed from baseline (defined as time point 1, before induction) until the end of the surgery and laryngeal mask removal (defined as time point 6). Data will be reported within one year after study completion
  • To assess the usefulness of general anesthesia with LMA-Classic for the endovascular treatment of cerebral aneurysms based on cardiovascular stability analysis

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Gomez Oquendo, MD, Principal Investigator — Department of Anesthesiology, University of Antioquia, Medellin, Colombia.

IPD SHARING:
Plan to Share IPD: No
De-identified data will be shared with our colleagues at The Ohio State University for posterior data analysis

REFERENCES:
- [Background] Brown RD Jr, Broderick JP. Unruptured intracranial aneurysms: epidemiology, natural history, management options, and familial screening. Lancet Neurol. 2014 Apr;13(4):393-404. doi: 10.1016/S1474-4422(14)70015-8. PMID 24646873
- [Background] Brisman JL, Song JK, Newell DW. Cerebral aneurysms. N Engl J Med. 2006 Aug 31;355(9):928-39. doi: 10.1056/NEJMra052760. No abstract available. PMID 16943405
- [Background] Weir B, Disney L, Karrison T. Sizes of ruptured and unruptured aneurysms in relation to their sites and the ages of patients. J Neurosurg. 2002 Jan;96(1):64-70. doi: 10.3171/jns.2002.96.1.0064. PMID 11794606
- [Background] Chowdhury T, Cappellani RB, Sandu N, Schaller B, Daya J. Perioperative variables contributing to the rupture of intracranial aneurysm: an update. ScientificWorldJournal. 2013 Nov 12;2013:396404. doi: 10.1155/2013/396404. PMID 24324371
- [Result] Lee CZ, Young WL. Anesthesia for endovascular neurosurgery and interventional neuroradiology. Anesthesiol Clin. 2012 Jun;30(2):127-47. doi: 10.1016/j.anclin.2012.05.009. Epub 2012 Jul 13. PMID 22901603
- [Result] Kundra S, Mahendru V, Gupta V, Choudhary AK. Principles of neuroanesthesia in aneurysmal subarachnoid hemorrhage. J Anaesthesiol Clin Pharmacol. 2014 Jul;30(3):328-37. doi: 10.4103/0970-9185.137261. PMID 25190938